CLINICAL TRIAL: NCT02086903
Title: Pharmacodynamic Effect of Loading And Maintenance Doses Of Clopidogrel Versus Half Doses of Ticagrelor In Healthy Subjects
Brief Title: Clopidogrel And Ticagrelor in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, MD. Director, Regional Clinical Trial Center. Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: COLLATERAL
Record Dates: First submitted 2014-03-12; First posted 2014-03-13 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Pharmacodynamics
Keywords: Ticagrelor; Clopidogrel; Platelet function test
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor 90 mg (Experimental): The subjects administer Ticagrelor 90 mg as loading dose (LD) follow by 90 mg/day as maintenance dose (MD) for 5 days, following a 2-week washout period, to receive the alternate thienopyridine (Clopidogrel 600 mg as LD follow by 75 mg/day as MD for 5 days).
  Interventions: Drug: Ticagrelor 90 mg
- Clopidogrel 600 mg (Experimental): The subjects administer Clopidogrel 600 as loading dose (LD) follow by 75 mg/day as maintenance dose (MD) for 5 days, following a 2-week washout period, to receive the alternate thienopyridine (Ticagrelor 90 mg/day as LD, follow by 90 mg/day as MD for 5 days).
  Interventions: Drug: Clopidogrel 600 mg

INTERVENTIONS:
Drug: Ticagrelor 90 mg — The subjects administer Ticagrelor 90 mg as loading dose (LD) follow by 90 mg/day as maintenance dose (MD) for 5 days, following a 2-week washout period, to receive the alternate thienopyridine (Clopidogrel 600 mg as LD follow by 75 mg/day as MD for 5 days).
  Other Names: Brilinta 90 mg
  Arms: Ticagrelor 90 mg
Drug: Clopidogrel 600 mg — The subjects administer Clopidogrel 600 as loading dose (LD) follow by 75 mg/day as maintenance dose (MD) for 5 days, following a 2-week washout period, to receive the alternate thienopyridine (Ticagrelor 90 mg/day as LD, follow by 90 mg/day as MD for 5 days).
  Other Names: Plavix 600 mg
  Arms: Clopidogrel 600 mg

SUMMARY:
To evaluate the pharmacodynamics of a lower Ticagrelor dose in healthy Korean volunteers compared with standard Clopidogrel agent.

DETAILED DESCRIPTION:
Consist with previous study Ticagrelor had greater, faster and more the platelet inhibition effect than Clopidogrel in both healthy subjects and stable coronary artery disease patients. Moreover, Asian subjects exposed higher active metabolite and stronger pharmacodynamics response than European subjects with same oral dose of antiplatelet agent. However, previous report comparing the efficacy and safety of Ticagrelor and Clopidogrel in healthy Asian ethnicity is lacking. Therefore, the aim of this study is to evaluate the pharmacodynamic responses of a lower Ticagrelor dose using laboratory platelet function tests in healthy Korean volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 12 healthy men
* Aged between 19 and 59 years
* Body mass index (BMI) is between 18.5 and 29.9 kg/m2
* Baseline maximal platelet aggregation (MPA) 10 μmol/L ADP is more than 65%
* To screen for standard results on usual clinical tests

Exclusion Criteria:

* A history of bleeding within 6 months
* Bleeding diathesis
* Hemoglobin < 12g/dl
* History of antiplatelet or anticoagulation treatment within 1 month
* contraindication to the study drug
* Severe hepatic dysfunction (serum liver enzyme or bilirubin >3 times normal limit)
* Patients with hereditary disease such as galactose intolerance, lactase deficiency, glucose-galactose malabsorption
* Previous experience of clinical trials within three months

Ages: 19 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | up to 122 hours
  Platelet reactivity will be measured using multiple platelet function tests, including, light transmission aggregometry (LTA), multiple electrode platelet aggregometry (MEA, Dynabyte Medical, Munich, Germany), VerifyNow (Accumetrics, San Diego, CA, USA), Total thrombus-formation analysis system (T-TAS®, Fujimori Kogyo, Japan). The platelet reactivity will be measured at 0.5, 2, 6, 24,26,120,122 hours after study drug administration.
  Percent inhibition is calculated using the following formula: % inhibition =[(baseline reactivity unit - gain(t) reactivity unit) / baseline reactivity unit] × 100.
  * Baseline reactivity unit is the value before Ticagrelor or Clopidogrel loading dose.
  * Gain(t) reactivity unit is the value for each subject at selected time points ( 0.5, 2, 6, 24,26,120,122 hours after study drug administration).

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, M.D., Principal Investigator — Dong-A University Hospital, Busan, Republic of Korea
Locations (1):
- Dong A University Hospital, Busan, South Korea

REFERENCES:
- [Background] Teng R, Mitchell P, Butler K. Effect of age and gender on pharmacokinetics and pharmacodynamics of a single ticagrelor dose in healthy individuals. Eur J Clin Pharmacol. 2012 Aug;68(8):1175-82. doi: 10.1007/s00228-012-1227-4. Epub 2012 Feb 25. PMID 22367426
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Kim MH, Zhang HZ, Jung DK. Pharmacodynamic comparisons for single loading doses of prasugrel (30 mg) and clopidogrel (600 mg) in healthy Korean volunteers. Circ J. 2013;77(5):1253-9. doi: 10.1253/circj.cj-12-0783. Epub 2013 Jan 30. PMID 23363643